CLINICAL TRIAL: NCT03966586
Title: Syndemics and Loss from the HIV Care Continuum in India - Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: YR Gaitonde Centre for AIDS Research and Education (Other)
Responsible Party: Principal Investigator, Brian Chan, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019P001573
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2022-07

CONDITIONS: HIV Infections
Keywords: hiv; India; retention; continuum
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Appointments and Schedules; Financial Support; Small Business; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Care (Experimental): Usual clinical care + intervention components
  Interventions: Behavioral: Active outreach; Behavioral: Appointments; Behavioral: Financial support; Behavioral: Microenterprise; Behavioral: Enhanced counseling
- Usual Care (Active Comparator): Usual clinical care and counseling
  Interventions: Behavioral: Usual clinical care and counseling

INTERVENTIONS:
Behavioral: Active outreach — Participants will get bidirectional weekly SMS messaging / automated voice messaging (depending on literacy), with messages to be programmed by the participant in the enhanced counseling sessions.
  Arms: Enhanced Care
Behavioral: Appointments — Participants in the enhanced-care intervention will be given specific appointment times/dates.
  Arms: Enhanced Care
Behavioral: Financial support — Participants in the enhanced-care intervention will receive free clinic visits, labs, and medications. They will also receive transportation incentives on a sliding scale based on distance to clinic, to range between 200-700 INR to be given each clinic/study visit. All participants, in both the usual care and enhanced care arms, will be offered VL testing free of charge, although this will not be known to the participants prior to the visit.
  Arms: Enhanced Care
Behavioral: Microenterprise — YRG CARE is affiliated with two microenterprise programs in bag-making and food-vending which can be leveraged as part of an intervention, particularly for women. There is an established training and mentoring program for individuals who wish to join the bag-making or food-making ventures. Participants who opt for this will be linked to the bag-making and food-vending programs, with all up-front costs (e.g. vending kiosk, training, serving materials, etc.) covered.
  Arms: Enhanced Care
Behavioral: Enhanced counseling — Participants in the enhanced-care intervention will participant in an individual enhanced counseling program called Steps to Success, based upon a Life Steps and Problem Solving curriculum. Steps to Success will consist of five one-on-one sessions of approximately 1 to 1.5 hours each. The first session will take place at the time of the participant's second clinical visit to YRG CARE, which will be between 1-3 weeks after the participant is recruited.
  Arms: Enhanced Care
Behavioral: Usual clinical care and counseling — Usual clinical care and counseling
  Arms: Usual Care

SUMMARY:
The investigators will assess the feasibility and acceptability of a pilot intervention to keep people living with HIV (PLHIV) in southern India in care and virologically suppressed. The lack of understanding of the causes of loss from the HIV care continuum in India stifles the armamentarium of effective interventions to keep Indian PLHIV in care. The results of this research will demonstrate the feasibility and acceptability of a pilot intervention targeting the multiple mechanisms by which PLHIV become lost to care. By targeting these mechanisms, this intervention will be designed to be scalable in a setting where access to mental health specialists is limited.

DETAILED DESCRIPTION:
This pilot intervention represents the final Aim of the NIMH-sponsored study "Syndemics and Loss from the HIV Care Continuum in India." This trial will be conducted at the Y.R. Gaitonde Centre for AIDS Research and Education (YRG CARE), located in Chennai, the capital of Tamil Nadu state and one of the epicenters of the Indian HIV epidemic.

The investigators will recruit 50 adult (age >=18) PLHIV presenting to care at YRG CARE and ART-naïve. Participants will be recruited at their first visit to YRG CARE, at which the participant's HIV diagnosis is established or confirmed and the participant receives initial counseling and clinical care. At this recruitment stage, research assistants will conduct a pre-intervention questionnaire including measures of depressive symptoms, internalized stigma, self-efficacy, mental health, and physical health. The investigators will then randomize the patient to usual care vs. enhanced-care intervention (25 in each arm).

The enhanced-care intervention will be multi-faceted, reflecting the likelihood of multiple syndemic conditions as well as evidence from LMICs suggesting that programs combining multiple approaches are the most effective in improving retention in care.

The enhanced-care intervention will consist of the following components:

1. Active outreach, including bidirectional weekly SMS messaging / automated voice messaging (depending on literacy)
2. Appointments (specific appointment times/dates).
3. Financial support, including free clinic visits, labs, medications, and transportation incentives on a sliding scale based on distance to clinic
4. Microenterprise, including bag-making or food-making ventures for women
5. Enhanced counseling. Participants in the enhanced-care intervention will participate in an individual enhanced counseling program called Steps to Success, based upon a Life Steps and Problem Solving curriculum.

ELIGIBILITY:
Inclusion Criteria:

* Adult PLHIV presenting to care at YRG CARE who are ART-naïve and who plan to follow-up at YRG CARE
* Speaks Tamil, Telugu, or English

Exclusion Criteria:

* Previous ART exposure
* Not competent to provide informed consent or participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by semi-structured qualitative interviews | 12 months
  Minimal negative impact on clinical work flow and ability to deliver all intervention components, particularly all sessions of enhanced counseling, as measured by semi-structured qualitative interviews of providers
Acceptability among participants and providers as assessed by semi-structured qualitative interviews | 12 months
  Acceptability among patients and providers as measured by semi-structured qualitative interviews of participants and providers

SECONDARY OUTCOMES:
Retention in care | 12 months
  No unexpected absences > 90 days
Viral suppression (Undetectable HIV-1 RNA, <50 copies / mL) | 3 months
  Undetectable HIV-1 RNA, <50 copies / mL
ART initiation success (accepted ART and continued ART for at least 6 months) | 6 months
  Successful ART initiation (accepted ART and continued ART for at least 6 months)
Depressive symptoms as measured by PHQ-9 | 12 months
  Score of >10 indicates probable depression
Internalized stigma as measured by Internalized AIDS-Related Stigma Scale | 12 months
  Includes six items related to concerns about disclosure as well as items related to feelings of shame and/or self-hatred. Responses are elicited on a binary scale (yes/no) and scores represent the sum of endorsed items.
Self-efficacy as measured by General Self-Efficacy Scale--shortened version | 12 months
  Six item scale of self-efficacy
Social support as measured by Multidimensional Scale of Perceived Social Support | 12 months
  12 item scale of social support
Food insecurity as measured by Household Food Insecurity Access Scale | 12 months
  8 item scale of food insecurity

CONTACTS AND LOCATIONS:
Locations (1):
- YRG CARE, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No